CLINICAL TRIAL: NCT02561546
Title: A Phase II Study to Investigate Preliminary Efficacy Using p53 Gene Therapy for Treatment of Diabetes Concurrent With Hepatocellular Carcinoma
Brief Title: p53 Gene Therapy in Treatment of Diabetes Concurrent With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: p53-DB-001
Record Dates: First submitted 2015-09-11; First posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-07

CONDITIONS: HCC; Diabetes
Keywords: concurrent
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAE plus p53 gene therapy (Experimental): Trans-catheter embolization (TAE) combined with recombinant adenoviral human p53 gene (rAd-p53) will be given one per month
  Interventions: Drug: p53 gene therapy; Drug: Trans-catheter embolization
- Trans-catheter embolization (Active Comparator): Trans-catheter embolization (TAE) will be given once per month
  Interventions: Drug: Trans-catheter embolization

INTERVENTIONS:
Drug: p53 gene therapy — Trans-catheter embolization (TAE) combined with recombinant adenoviral human p53 gene (rAd-p53) will be given one per month
  Other Names: recombinant adenoviral human p53 gene therapy
  Arms: TAE plus p53 gene therapy
Drug: Trans-catheter embolization — Trans-catheter embolization alone

SUMMARY:
An open-labeled phase II study to investigate preliminary efficacy using p53 gene therapy in treatment of diabetes concurrent with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
It was found in the treatment of HCC using p53 gene therapy that the concurrent diabetes was controlled as well. The objectives of this study are to investigate both anti-diabetic and anti-tumor role of p53 gene therapy. This is an open-labeled, randomized, active-controlled phase 2 study. p53 will be injected via the artery, which supplies blood for the tumor nodules. The study endpoints for anti-diabetic role are fasting plasma glucose (FPG), postprandial glucose (PPG) and glycosylated hemoglobin (A1C) at 30 days after the start of treatment; and for antitumor effect are progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically diagnosed unresectable HCC
* over 18 years old
* with an Eastern Cooperative Oncology Group (ECOG) score of 0-2
* with Barcelona Clinic Liver Cancer (BCLC) Stage of B or C
* with Child-Pugh score A or B; with normal tests of hemogram, blood coagulation, liver and kidney function
* signed the informed consent form.

Exclusion Criteria:

* hypersensitive to study drug
* With an abnormal coagulation condition or bleeding disorder
* infections
* with serious conditions which prevent using the study treatment
* pregnant or lactating

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
fasting plasma glucose (FPG) | from starting treatment until 60 days
  In 60 days after starting study treatment
glycosylated hemoglobin (A1C) | from starting treatment until 60 days
  In 60 days after starting study treatment

SECONDARY OUTCOMES:
overall survival (OS) | 2 years
  overall survival will be follow up to 2 years. Time to an event (death), or censored status (lost of follow up, withdrawal from the study, or still alive on 2 years) will be recorded. OS will be estimated using Kaplan-Meier method.
progression free survival (PFS) | 2 years
  PFS will be follow up to 2 years. Time to an event (progression or death) or censored status (lost of follow up, withdrawal from the study, or still alive and no progression on 2 years). Assessment of progression will follow RECIST standard Version 1.1. PFS will be estimated using Kaplan-Meier method.
postprandial glucose (PPG) | from starting treatment until 60 days
  from starting treatment until 60 days treatment

CONTACTS AND LOCATIONS:
Locations (1):
- first affiliated hospital in Dalian University, Dalian, Liaoning, China